CLINICAL TRIAL: NCT04710199
Title: Proof-of-concept Trial to Evaluate the Safety and Efficacy of Maraviroc in Severe Acute Respiratory Syndrome (SARS) Coronavirus-2 (CoV-2) Infected Patients Hospitalized for COVID-19
Brief Title: Trial to Evaluate the Safety and Efficacy of Maraviroc in Patients Hospitalized for Coronavirus Disease 2019 (COVID-19)
Acronym: COVIMAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVIMAR
Record Dates: First submitted 2021-01-05; First posted 2021-01-14 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Virus Diseases
Keywords: Sar-COv19; coronavirus; COVID19
MeSH Terms: conditions — Virus Diseases; Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: In this clinical trial, standard treatment together with Maraviroc (MVC) is evaluated compared to treatment alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maraviroc experimental group (Experimental): Maraviroc tablet combined with standard treatment
  Interventions: Drug: Maraviroc experimental group
- Standard treatment (Other): It is based on the treatment protocol for hospitalized COVID-19 patients and that will depend on the clinical status of the patient.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: Maraviroc experimental group — 300-milligram dose of the drug two times daily , oral way. During 14 days.
  Arms: Maraviroc experimental group
Other: Standard treatment — It is based on the treatment protocol for hospitalized COVID-19 patients and that will depend on the clinical status of the patient.
  Arms: Standard treatment

SUMMARY:
Maraviroc (MVC) is a drug, very well tolerated, it has been seen that MVC has properties of modulating the immune system, exerting an anti-inflammatory effect in different diseases. In COVID-19, very high levels of inflammation occur that cause organs and systems to be damaged. MVC could reduce this inflammation achieving a better prognosis of COVID-19.

DETAILED DESCRIPTION:
In this clinical trial the investigators want to evaluate if standard treatment together with Maraviroc (MVC) compared to standard treatment alone, achieves better clinical evolution in participants hospitalized for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Infection confirmed by SARS-CoV-2 by polymerase chain reaction (PCR) at least 3 days before randomization.
* Hospitalized or emergency patient in hospitalization phase.
* Mild / moderate pneumonia, with fever, persistent cough and severe asthenia, confirmed by imaging tests (conventional radiology or computerized axial tomography (CT)) with ambient air oxygen saturation (SatO2)> 94%.
* Less than 12 days from the onset of symptoms.
* Women of childbearing potential must have a negative serum or urine pregnancy test prior to inclusion in the study and must commit to using highly effective contraceptive methods (intrauterine device, bilateral tubal occlusion, vasectomized partner, and sexual abstinence).
* Accepts written consent or oral informed in the case that due to the relevant security protocols, written consent is not possible.

Exclusion Criteria:

* Patient with severe pneumonia confirmed by imaging test (conventional radiology or computerized axial tomography (CT)) with ambient air oxygen saturation (SatO2) ≤94%.
* Another acute active infection other than that produced by SARS-CoV-2.
* Chronic renal failure (estimated glomerular filtration ≤ 30 ml / min / 1.73 m2 or receiving renal replacement therapy in any of its modalities).
* Known HIV infection. Unless the patient has> 500 CD4 + / mm3 and an undetectable viral load for more than 6 months.
* Active co-infection with known hepatitis B or C viruses.
* Cirrhosis, portal hypertension and / or hypersplenism of any etiology.
* Past or current neoplasms subsidiary to treatment with steroids, immunomodulators or chemotherapy
* Laboratory abnormalities.
* Concomitant use of drugs with major pharmacological interactions with the study drugs, according to the respective technical specifications of the products.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of Maraviroc in SARS-CoV-2 infected patients hospitalized for COVID-19 using the Ordinal scale. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Ordinal scale: (1) Not hospitalized, without limitations in activities; (2) Not hospitalized, limitations in activities; (3) Hospitalized, with no oxygen supplement requirement; (4) Hospitalized, requiring supplemental oxygen; (5) Hospitalized, with non-invasive ventilation or high flow oxygen device or oxygen mask with reservoir); (6) Hospitalized, with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); (7) Death. treatment versus standard treatment, in relation to the clinical progression of COVID-19 in hospitalized patients.

SECONDARY OUTCOMES:
Analyze changes in analytical variables: changes in ambient air oxygen saturation (SatO2),related to the progression of COVID-19. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Analytical variables related to the progression of COVID-19: changes in ambient air oxygen saturation (SatO2) (mmHg).
Study the variation in the number of biomarkers of inflammation. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels of macrophage inflammatory proteins-1 α (MIP-1 α), MIP-1 β, regulated on activation normal T cell expressed and secreted (RANTES), interleukin-6 (IL-6), IL-8, interferon-inducible protein 10 (IP-10), IL-1β, TNF-α, gamma interferon (IFN-γ), soluble cluster of differentiation 25 (CD25), β2 microglobulin, dimers D, soluble cluster of differentiation 14 (CD14), soluble cluster of differentiation 40 (CD40) ligand and soluble cluster of differentiation 163 (CD163).
Analyze changes in the number of innate immune activation (monocytes and dendritic cells) and adaptive (T lymphocytes). | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels subpopulations (classical, intermediate and non-classical monocytes) and activation markers in them. Dendritic cell subpopulations (myeloid and plasmacytoid dendritic cells) and their activation markers. Subpopulations of T lymphocytes (naive, central memory, effector memory and terminally differentiated) and markers of activation, senescence and wasting in them.
Quantify the number of immunomodulatory treatments added to therapy | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Quantification of additional treatments added to the administered therapy , this is immunomodulatory treatments such as: IL-6,or IL-1 inhibitors, high-dose corticosteroids, anti-tumor necrosis factor (anti-TNF) antibodies, janus kinases (JAK) kinase inhibitors or any other immunomodulatory effect and / or under investigation
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Analyze changes in analytical variables:changes in neutrophils, related to the progression of COVID-19. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels of neutrophils in blood (x10e9/L)
Analyze changes in analytical variables: changes in platelets, related to the progression of COVID-19. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels of platelets in blood (x10e9/L)
Analytical variables related to the progression of COVID-19: changes in lactate dehydrogenase (LDH). | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels of lactate dehydrogenase in blood (U/L)
Analyze changes in analytical variables: changes in C-reactive protein, related to the progression of COVID-19. | Baseline, change from baseline at 7 days, change from baseline at 14 days, change from baseline at 21 days and change from baseline at 28 days
  Changes in levels of C-reactive protein in blood (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Lomas, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen del Rocío, Seville